CLINICAL TRIAL: NCT01053390
Title: A Phase III Study of New Chemotherapy Regimen in the Treatment of Advanced Gallbladder Carcinoma
Brief Title: New Chemotherapy Regimen in the Treatment of Advanced Gallbladder Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Capital Medical University (Other); Peking University First Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); China Medical University, China (Other); The first clinical college of harbin medical university (Unknown); The Second Affiliated Hospital of Harbin Medical University (Other); Shengjing Hospital (Other); Jilin University (Other); The people's hospital of Heilongjiang province (Unknown); Eastern Hepatobiliary Surgery Hospital (Other); Shanghai Changzheng Hospital (Other); Shandong Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other); Air Force Military Medical University, China (Other); Tang-Du Hospital (Other); Qinghai People's Hospital (Other); Affiliated Hospital of Qinghai University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); First People's Hospital of Kunming (Other); Lanzhou University Second Hospital (Other); Xi'an Central Hospital (Other); The first people's hospital of Guiyang (Unknown); Southwest Hospital, China (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Zhi-wei Quan, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xh2009-35
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Gallbladder Neoplasms
Keywords: gallbladder neoplasmas; Gallbladder Neoplasms,Advanced Stage,Chemotherapy,Somatostatin
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Somatostatin; Epirubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epirubicin,cisplatin,LV（Leucovorin）、5-FU (5-Fluorouracil) (Active Comparator): conventional regimen
  Interventions: Drug: epirubicin, cisplatin, LV（Leucovorin）、 5-FU（5-Fluorouracil）
- Somatotatin (Experimental): Conventional chemotherapy regimen plus somatostatin
  Interventions: Drug: Somatostatin; Drug: epirubicin, cisplatin, LV（Leucovorin）、 5-FU（5-Fluorouracil）

INTERVENTIONS:
Drug: Somatostatin — Somatostatin 3mg+NS（normal saline）60ml, a continuous intravenous infusion, q12h
  Arms: Somatotatin
Drug: epirubicin, cisplatin, LV（Leucovorin）、 5-FU（5-Fluorouracil）

SUMMARY:
Objective Primary:

Determine the objective response rate in patients with advanced gallbladder treated with new Chemotherapy regimen

Secondary:

Determine time to progression-free survival and overall survival of patients treated with this regimen.

Determine quality of life of patients treated with this regimen. Determine the toxicity of new chemotherapy regimen

DETAILED DESCRIPTION:
Study Design: Treatment, Randomized, Open Label, controlled,Multicenter Group Assignment, Safety/Efficacy Study

Chemotherapy regimen:

Group A: Conventional chemotherapy regimen Group B: New chemotherapy regimen: conventional regimen plus SST（somatostatin） Cycles repeat every 4 weeks and 6 cycles in total

Patients: A total of 260 patients (130 per group) will be accrued for this study.

Patients distribution:

10patients per center are enrolled in the study and 30 centers (hospitals) in total which meet the total number of patients in trial.

Clinical Outcome Assessments:

Primary: the objective response rate (response evaluation criteria in solid tumors ,RECIST criteria) Secondary: progression-free survival, overall survival, quality of life，the adverse event

Safety Assessments:

Physical exam, laboratory test, probably occurred adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable locally advanced disease or unresectable local recurrence, including:

   * Patients with unresectable advanced gallbladder cancer （≥ Nevin staging IV or TNM（ tumor node metastasis） classification）
   * Patients with complication who have no indication for surgery
   * Patients with unresectable local recurrence lesions
2. Age between 18-75, no gender-based constraints
3. Estimated life expectancy ≥12 weeks
4. KPS（Karnofsky performance status ）≥60
5. Each patient gave written informed consent
6. < 2 previous chemotherapy regimes
7. No chemotherapy done in the last 4 weeks
8. Laboratory test criteria:Haemoglobin ≥ 10g/dl, white blood cell count > 3,000/mm3 ;Platelet >100,000/mm3 Total bilirubin <5.0mg/dl ALT（alanine transaminase）、 AST（aspartate aminotransferase)≤ 2.5 times upper limit of normal BUN（blood urea nitrogen）≤ 2 times upper limit of normal; serum creatinine <1.5mg/dl: creatinine clearance rate < 60 ml/min
9. Patients are required to have histologically confirmed diagnosis via puncture based at least on computed tomography (CT) or ultrasound
10. Jaundice should be reduced to standard level before chemotherapy (Total bilirubin <5.0 mg/dl)

Exclusion Criteria:

1. Patients with extensive metastasis and generally poor condition who can not tolerate chemotherapy
2. Patients who are pregnant or breastfeeding.
3. Patients with other clinically significant laboratory abnormalities, uncontrolled infection, concurrent severe medical problems unrelated to malignancy
4. Patients who had a history of previous carcinoma in the last 5 years.
5. Patients who are allergic to somatostatin or fluorouracil
6. Patients who refuse chemotherapy, or to sign the informed consent and chemotherapy consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
(Response Evaluation Criteria in Solid Tumors, RECIST,2009 ), CR(complete response) and PR(partial response) | 6 month after first treatment

SECONDARY OUTCOMES:
A: KPS (karnofsky performance score) B:Laboratory tests: Reexamination of CA19-9（Carbohydrate Antigen 19-9）、 CEA（ carcinoembryonic antigen）, especially for those which are abnormal prior to chemotherapy | 6 month after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-wei Quan, MD, Study Chair — Xinhua hospital affiliated shanghai jiaotong university school of medicine
Locations (1):
- Xinhua hospital affiliated shanghai jiaotong, Shanghai, China